CLINICAL TRIAL: NCT01243853
Title: Alpha-galactosidase Enzyme and Irritable Bowel Syndrome
Acronym: ALFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Verman Oy Ab (Industry)
Responsible Party: Jari Koskenpato/Principal Investigator, Gastrolääkärit Oy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: VER001
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — alpha-Galactosidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alpha-galactosidase (Active Comparator)
  Interventions: Dietary Supplement: Alpha-galactosidase
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Alpha-galactosidase

INTERVENTIONS:
Dietary Supplement: Alpha-galactosidase — 3 months intervention, daily 3 x 3 capsules alpha-galactosidase enzyme (400 GalU/capsule) or 3 x 3 capsules placebo

SUMMARY:
The purpose of this study is to determine whether alpha-galactosidase enzyme is affective in alleviating the symptoms of irritable bowel syndrome (IBS).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IBS according to Rome III criteria, additionally abdominal distension or flatulence the most disturbing symptom
* Age 18-65 years
* Colonoscopy conducted within the previous 5 years, finding macroscopically and histologically normal

Exclusion Criteria:

* Organic GI disease. Treated (min. 1 year) coeliac disease patients, and subjects with known and treated lactose intolerance are allowed to participate
* Malignancy
* Significant gastrointestinal surgery
* Clinically significant aberrancies in the screening-phase laboratory analyses
* Changes in regular medication during the previous 4 weeks
* Pregnancy or breast feeding
* Other disease or state that based on the investigator's evaluation complicates the conduction of the intervention, i.e. alcoholism, dementia
* Hereditary galactosemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
IBS symptom severity | baseline
  The IBS symptom severity score (IBS-SSS) questionnaire is used
IBS symptom severity | 1 month
  The IBS symptom severity score (IBS-SSS) questionnaire is used
IBS symptom severity | 2 months
  The IBS symptom severity score (IBS-SSS) questionnaire is used
IBS symptom severity | 3 months
  The IBS symptom severity score (IBS-SSS) questionnaire is used
IBS symptom severity | follow-up (4 months)
  The IBS symptom severity score (IBS-SSS) questionnaire is used

CONTACTS AND LOCATIONS:
Overall Officials: Jari Koskenpato, MD, PhD, Principal Investigator — Gastrolääkärit Oy
Locations (1):
- Gastrolääkärit Oy, Helsinki, Finland